CLINICAL TRIAL: NCT07312149
Title: BoxTer : Isolation of Pulmonary Veins Using the Box Technique in Patients Undergoing Sternotomy
Brief Title: Isolation of Pulmonary Veins Using the Box Technique in Patients Undergoing Sternotomy
Acronym: BoxTer
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC25_0420
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Cardiac Surgery
Keywords: Atrial firbrillation; Cardiac Surgery; PWI-Box; GeminiS
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BOXTER Study population: Patients with a surgical indication for AF in combination with conventional cardiac surgery performed by sternotomy (coronary artery bypass grafting, aortic valve replacement, aortic surgery, etc.).
  Interventions: Other: Collection of study data from patient records

INTERVENTIONS:
Other: Collection of study data from patient records — Collection of study data from patient records in the EPICARD national database at the time of surgery, 1 month post-surgery, 12 months post-surgery, 24 months post-surgery and 36 months post-surgery.

SUMMARY:
Atrial Fibrillation (AF) is the most common cardiac arrhythmia worldwide, affecting approximately 2.8% of the population, with prevalence increasing with age. AF is associated with significant morbidity and mortality, accounting for about 25% of ischemic strokes, 10% of cryptogenic strokes, and a 10-40% annual increase in hospital admissions due to heart failure or anticoagulant-related events.

About 10% of patients undergoing cardiac surgery have preoperative AF. In 1986, Dr. Cox introduced the MAZE procedure, a surgical technique to isolate AF triggers. Initially involving atrial incisions, it evolved to use radiofrequency lines, significantly reducing morbidity and mortality. The MAZE procedure is now strongly recommended (Class Ia evidence) for concomitant cardiac surgery. However, nearly 85% of eligible patients-especially those undergoing closed-chest cardiac surgery-do not receive this treatment due to technical challenges and limited reproducibility of the Cox-Maze IV technique.

Pulmonary Vein Isolation (PVI) with posterior wall isolation (PWI-Box) has emerged as an effective alternative, offering similar outcomes to Cox-Maze IV with fewer adverse effects. Innovative devices like the GeminiS (Medtronic) enable minimally invasive, thoracoscopic PVI-PWI-Box procedures without opening the heart, even off-pump. This approach could expand the use of AF ablation during combined sternotomy surgeries, aligning with clinical guidelines.

Primary Objective: Assess the efficacy of PWI-Box using GeminiS combined with other cardiac surgeries via sternotomy.

Primary Endpoint: Recurrence rate of paroxysmal or persistent AF (per ESC definition) at 1 year postoperatively, confirmed by 24-hour Holter monitoring.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing cardiac surgery via sternotomy
* Concomitant use of the PWI box with GeminiS during surgery
* Adult patients
* Patients with the following characteristics: Preoperative paroxysmal/persistent/permanent AF; Duration of less than 5 years; And left atrium volume <60 ml/m2
* Informed patient who did not object to the collection of their data for the study

Exclusion criteria:

* Unplanned surgery (emergency)
* History of cardiac surgery (reoperation)
* Pregnant or breastfeeding women
* Adults under guardianship, curatorship or judicial protection
* Patients with a life expectancy of less than three years
* Patients currently taking medication or using an experimental device that clinically interferes with the study's evaluation criteria and results.
* Inability to comply with the monitoring schedule.
* Contraindication to long-term anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a surgical indication for AF in combination with conventional cardiac surgery performed by sternotomy (coronary artery bypass grafting, aortic valve replacement, aortic surgery, etc.). Patients may be included prospectively, via information provided by the attending physician during a consultation (written and oral), or retrospectively for those who have already undergone surgery, by sending an information notice with a non-objection period.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2030-01-05 (Estimated); Study Completion 2032-01-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of the PWI box, using GeminiS in combination with other cardiac surgery procedures via sternotomy, at 1 year post-operatively using 24-hour Holter monitoring. | 12 months

SECONDARY OUTCOMES:
Evaluation of the efficacy of the PWI box using GeminiS in combination with other cardiac surgery procedures via sternotomy at 2 years postoperatively. | 24 months
Evaluation of the efficacy of the PWI box using GeminiS in combination with other cardiac surgery procedures via sternotomy at 3 years postoperatively. | 36 months
Evaluation of the rate of secondary endocardial ablation of AF. | 12 months
Evaluation of clinicals predictive factors for recurrence of AF after MAZE. | 36 months
Evaluate the rate of patients on anticoagulant and/or antiarrhythmic therapy after MAZE surgery. | 36 months
Assessment of complication rates associated with the technique used during cardiac surgery. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Henri DAVID, Study Director — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided